CLINICAL TRIAL: NCT00942409
Title: A Phase II Study of Repeat Intranodal Injections of Adenovirus-CD154 (Ad-ISF35) in Patients With Non-Hodgkin's Lymphoma (Follicular, Diffuse Large Cell, Mantle Cell and Small Lymphocytic Lymphoma/Chronic Lymphocytic Leukemia)
Brief Title: Study of Repeat Intranodal Injections of Ad-ISF35
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: drug supply was no longer available
Sponsor: Januario Castro, M.D. (Other)
Collaborators: Memgen, LLC (Industry)
Responsible Party: Sponsor-Investigator, Januario Castro, M.D., Associate Clinical Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSD-101358 - prev 081503
Record Dates: First submitted 2009-07-17; First posted 2009-07-20 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-11

CONDITIONS: Non-Hodgkin's Lymphoma; Follicular Lymphoma; Diffuse Large Cell Lymphoma; Mantle Cell Lymphoma; Small Lymphocytic Lymphoma; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ad-ISF35 (Experimental): Ad-ISF35, intranodal injection, 3.3 x 10^10 ISF35 viral particles, every 2-4 weeks up to six total injections.
  Interventions: Biological: ISF35

INTERVENTIONS:
Biological: ISF35 — Subjects participating in this study will be treated with multiple doses of Ad-ISF35 given via intranodal injection using a fixed dose of 3.3 x 10^10 ISF35 viral particles. Intranodal injections will be administered every 2-4 weeks up to six total injections.

SUMMARY:
This is a Phase II, open label, fixed dose, repeat injection, single institution study. Eligible subjects will receive up to six doses of Ad-ISF35 injected directly into a selected lymph node under ultrasound guidance. The primary goal is to determine and monitor clinical and biological responses in patients treated with repeat intranodal injections of Ad-ISF35.

DETAILED DESCRIPTION:
This is a phase II clinical trial in which study subjects will be treated with multiple doses of Ad-ISF35 given via intranodal injection using a fixed dose of 3.3 x 10^10 ISF35 viral particles. Intranodal injections will be administered every 2-4 weeks up to six total injections.

This will be the first time that repeat administration of Ad-ISF35 will be performed via intranodal injection in subjects with a diagnosis other than CLL/SLL. Therefore, in order to allow sufficient time to evaluate the safety and toxicity of this procedure in non-CLL/SLL patients, we will treat the first three non-CLL/SLL subjects with inpatient admission for 24 hours observation at the GCRC-UCSD. If no serious adverse events are observed in these first three patients after they have received their first two injections of ISF35 and have been observed for at least 28 days, then we will proceed with enrollment of cohorts of four subjects per month. This will be done at one week intervals until study enrollment is completed. These subjects will be treated as outpatients at the GCRC and observed for 3 hours prior to discharge.

All subjects with a diagnosis of CLL or SLL will be treated as outpatients at the GCRC and observed for 3 hours prior to discharge. These subjects will not need to be treated in an inpatient setting, based on our previous clinical experience with subjects enrolled on the phase II study of repeat intranodal injections of Ad-ISF35 in CLL/SLL

ISF35 has already been used in Phase I clinical trials. The trials demonstrated that ISF35 treatment is well-tolerated and patients did not experience any significant or unexpected adverse events. Patients reported flu-like symptoms from ISF35, which disappeared within one to three days.

ISF35 is an abbreviation for Immune Stimulatory Factor 35, an offspring of technology discovered by Dr. Thomas J. Kipps, MD, PhD, Professor, Department of Medicine and Deputy Director for Research,UCSD Moores Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

SLL / CLL PATIENTS

1. Diagnosis of B-cell SLL/ CLL including

   * Lymphocytosis of monoclonal B-cells co-expressing ≥ one B-cell marker (CD19, CD20, or CD23) and CD5 in peripheral blood or lymph node AND
   * Bone marrow with ≥ 30% mononuclear cells having the SLL / CLL phenotype.
2. Presence of at least ONE single accessible AND palpable lymph node in the cervical, supraclavicular, axillary, or inguinal regions. The size of the lymph nodes must be larger than 2x2 cm in the horizontal and perpendicular axes.
3. Intermediate or High risk, poor prognosis SLL / CLL
4. Indication for treatment as defined by the NCI Working Group Guidelines:

   * Massive (i.e. > 6 cm below the left costal margin) or progressive splenomegaly OR
   * Massive lymph nodes or nodal clusters (i.e. > 10 cm in longest diameter), or progressive lymphadenopathy OR
   * Grade 2 or 3 fatigue OR
   * Fever ≥ 100.5˚F or night sweats for greater than 2 weeks without documented infection OR
   * Presence of weight loss ≥ 10% over the preceding 6 months OR
   * Progressive lymphocytosis with an increase of ≥ 50% over a 2-month period or an anticipated doubling time of less than 6 months.
   * Evidence of progressive marrow failure as manifested by the development of, or worsening of, anemia and / or thrombocytopenia.
   * Autoimmune anemia and / or thrombocytopenia poorly responsive to corticosteroid therapy.

   NHL PATIENTS
5. Non-Hodgkin's Lymphoma patients that have received at least one prior treatment (Antibodies and / or chemotherapy). Patients must have one of the following subtypes according to the WHO/REAL Classification[1]: follicular lymphoma, diffuse large cell lymphoma, mantle cell lymphoma and small lymphocytic lymphoma / chronic lymphocytic lymphoma.
6. Stage III or IV disease at any time in the past (Ann Arbor Staging System for Non-Hodgkin's Lymphomas).
7. Presence of at least ONE single accessible AND palpable lymph node in the cervical, supraclavicular, axillary, or inguinal regions. The size of the lymph nodes must be larger than 2x2 cm in the horizontal and perpendicular axes.

   ALL PATIENTS
8. Males and females 18 years of age and older
9. Laboratory parameters as specified below:

   * Hematologic: Hemoglobin ≥ 10 g/dL (may be post-transfusion); platelet count ≥ 50 x103/mm3
   * Hepatic: Total Bilirubin < 2 X ULN, and ALT and AST < 2 x ULN
   * Renal: Creatinine ≤ 2 X ULN
10. ECOG Performance Status ≤ 2
11. Anticipated survival of at least 3 months
12. For men and women of child-producing potential, use of effective barrier contraceptive methods during the study and for one month following treatment.
13. Ability to understand the requirements of the study, provide written informed consent and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and return for the required assessments.
14. Negative test results for current/active infection with HIV-1, HIV-2, HTV-1, HTLV-2, hepatitis A, B, C within 30 days of registration. (Antibody, antigen and nucleic acid tests acceptable, depending on institutional standards.).
15. Subjects must give written informed consent to participate in this trial.

Exclusion Criteria:

1. Pregnant or nursing women
2. Treatment with chemotherapy or monoclonal antibody within 28 days prior to entering the study.
3. Treatment with chemotherapy or monoclonal antibody during the time of participation in this trial.
4. Grade 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification
5. Severe or debilitating pulmonary disease (dyspnea at rest, significant shortness of breath, COPD).
6. Participation in any investigational drug study within 28 days prior to ISF35 administration. (Patient must have recovered from all acute effects of previously administered investigational agents).
7. Evidence of aggressive or highly aggressive lymphoma or Richter's transformation based on WHO/REAL classification criteria[1]
8. Any T cell lymphoma.
9. History of malignancy other than NHL or SLL/CLL or within five years of registration, except patients with adequately treated basal, squamous cell carcinoma or localized cervical cancer.
10. Active symptomatic fungal, bacterial and/or viral infection including active HIV or viral (A, B or C) hepatitis.
11. Any illness or condition that in the opinion of the Investigator may affect safety of treatment or evaluation of any the study's endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Januario Castro, M.D., Principal Investigator — Associate Clinical Professor in the Blood and Bone Marrow Transplantation Division; Thomas J Kipps, M.D., Ph.D., Principal Investigator — Professor of Medicine, Evelyn and Edwin Tasch Chair in Cancer Research in the UCSD School of Medicine
Locations (1):
- University of California, San Diego Moores Cancer Center, La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ad-ISF35
Started | 5
Completed | 2
Not Completed | 3
Not completed — Lack of Efficacy | 1
Not completed — study drug unavailable | 2

BASELINE CHARACTERISTICS:
Arm/Group | Ad-ISF35
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Time Frame: 2 Years
Population: The study was not completed due to unavailability of the study drug, and therefore data were not collected for this Outcome Measure
Arm/Group | Ad-ISF35
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Ad-ISF35
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ad-ISF35 (N=5)
Hyponatremia (General disorders) | 1
Anorexia/Early satiety (General disorders) | 5
Chills (General disorders) | 5
Fatigue (General disorders) | 5
Fever (General disorders) | 5
Flu like Syndrome (Immune system disorders) | 5
Injection site reaction (Immune system disorders) | 5
Nausea (Gastrointestinal disorders) | 5
Sweating (General disorders) | 5
Vomiting (Gastrointestinal disorders) | 4
Weight loss (General disorders) | 4
Cough (General disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Hematuria (Renal and urinary disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes